CLINICAL TRIAL: NCT01578239
Title: A Multicentre, Stratified, Open, Randomized, Comparator-controlled, Parallel-group Phase III Study Comparing Treatment With 177Lu-DOTA0-Tyr3-Octreotate to Octreotide LAR in Patients With Inoperable, Progressive, Somatostatin Receptor Positive Midgut Carcinoid Tumours
Brief Title: A Study Comparing Treatment With 177Lu-DOTA0-Tyr3-Octreotate to Octreotide LAR in Patients With Inoperable, Progressive, Somatostatin Receptor Positive Midgut Carcinoid Tumours
Acronym: NETTER-1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Advanced Accelerator Applications (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AAA-III-01; 2011-005049-11 (EudraCT Number); CAAA601A12301 (Other: Novartis)
Record Dates: First submitted 2012-04-10; First posted 2012-04-16 (Estimated); Results first posted 2017-10-02 (Actual); Last update posted 2022-04-04 (Actual); Status verified 2022-02

CONDITIONS: Carcinoid Tumor of the Small Bowel; Neuroendocrine Tumour
Keywords: Neuroendocrine tumour; 177Lu-Dota0-Tyr3-octreotate
MeSH Terms: conditions — Neuroendocrine Tumors | interventions — Octreotide; lutetium Lu 177 dotatate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 177Lu-DOTA0-Tyr3-Octreotate (Experimental): * 30 mg Octreotide LAR treatment for symptom control continued until the end of study, unless the participant progressed or died.
  * Treatment consisted of a cumulative administered radioactivity of 29.6 Giga Becquerel (GBq) (800 mCi) 177Lu-DOTA0-Tyr3-Octreotate: Four administrations of 7.4 GBq (200 mCi).
  * Concomitant amino acids were given with each administration for kidney protection.
  * 177Lu-DOTA0-Tyr3-Octreotate was administered at 8 +/- 1-week intervals, which could be extended up to 16 weeks to accommodate resolving acute toxicity.
  * In case participants experienced clinical symptoms (i.e. diarrhoea and flushing) associated with their carcinoid tumours, Octreotide s.c. rescue injections were allowed.
  Interventions: Drug: Octreotide LAR; Drug: 177Lu-DOTA0-Tyr3-Octreotate
- Octreotide LAR (Active Comparator): * 60 mg Octreotide LAR treatment every 4 weeks (i.m. injections) until the end of the study, unless the participant progressed or died.
  * In case participants experienced clinical symptoms (i.e. diarrhoea and flushing) associated with their carcinoid tumours, s.c. Octreotide rescue injections were allowed.
  Interventions: Drug: Octreotide LAR

INTERVENTIONS:
Drug: Octreotide LAR — In the experimental arm, 30 mg Octreotide LAR treatment was given to the participants until the end of study for symptom control purpose, unless the participant progressed or died.
  In the active comparator arm, 60 mg Octreotide LAR treatment was given to the participants every 4 weeks (i.m. injections) until the end of the study, unless the participant progressed or died.
  Other Names: SANDOSTATIN LAR, Octreotide
Drug: 177Lu-DOTA0-Tyr3-Octreotate — Four administrations of 7.4 GBq (200 mCi) 177Lu-DOTA0-Tyr3-Octreotate administered at 8 +/- 1-week intervals, which could be extended up to 16 weeks to accommodate resolving acute toxicity.
  Other Names: Lutathera
  Arms: 177Lu-DOTA0-Tyr3-Octreotate

SUMMARY:
This was a multicenter, stratified, open, randomized, comparator-controlled, parallel-group phase III study comparing treatment with Lutathera plus best supportive care (30 mg Octreotide LAR) to treatment with high dose (60 mg) Octreotide LAR in participants with metastasized or locally advanced, inoperable, somatostatin receptor positive, histologically proven midgut carcinoid tumours with progression despite LAR treatment.

DETAILED DESCRIPTION:
After the screening period, participants who signed the ICF and were eligible for the study in accordance with the entry criteria were randomly assigned to treatment either Lutathera or Octreotide LAR. Participant randomization was performed according to a centralized permuted block randomization scheme with a balanced ratio (1:1) between the 2 treatment groups, stratified by tumor uptake score and by the length of time that a participant was on a constant dose of Octreotide (=< 6 versus > 6 months).

Objective tumor assessment in both groups was performed every 12+/-1 weeks from the randomization date according to RECIST Criteria until progression was centrally confirmed:

1. Any participants with progressive disease (confirmed by central review of CT/MRI scans) ceased the treatment/assessment period and proceeded to the long-term follow-up period for evaluation of survival and long-term safety.
2. All non-progressive participants continued treatment/assessments until the PFS primary endpoint was met (i.e. 74 evaluable and centrally confirmed disease progressions or death events). Once the Primary End-Point was reached:

   1. Participants who received more than 76 weeks of treatment/assessment, stopped the study treatment (however somatostatin analogues could be received as subsequent treatment as per Investigator's discretion) but continued the long-term follow-up assessment for 5 years overall from the date of randomization of the last participant randomized.
   2. The remaining randomized participants continued in the fixed 76-week treatment/assessment period unless progression occurred, then continued the long-term follow-up assessments for 5 years overall from the date of randomization of the last participant.

ELIGIBILITY:
Inclusion Criteria:

1. Presence of metastasized or locally advanced, inoperable (curative intent) at enrollment time, histologically proven, midgut carcinoid tumour (to be centrally confirmed).
2. Ki67 index ≤ 20% (to be centrally confirmed).
3. Patients on Octreotide LAR at a fixed dose of 20 mg or 30 mg at 3-4 weeks intervals for at least 12 weeks prior to randomization in the study.
4. Patients ≥18 years of age.
5. Patients must have progressive disease based on RECIST Criteria, Version 1.1 while receiving an uninterrupted fixed dose of Octreotide LAR (20-30 mg/3-4 weeks). Disease progression must be centrally confirmed. In order to make the assessment, two CT (or MRI) scans are required. The oldest scan must not be older than 3 years from the date of randomization. The most recent scan must not be older than 4 weeks from the date of randomization. Both scans must be obtained while the patient is receiving the same fixed dose of Octreotide LAR (20-30 mg/3-4 weeks) with the following exceptions; 1) it is acceptable if the oldest scan is obtained within 12 weeks of the patient receiving a fixed dose regimen of Octreotide LAR (20-30 mg/3-4 weeks); AND 2) it is acceptable for either scan to be obtained before or during the time a patient receiving a fixed dose of Octreotide LAR has switched to an equivalent dose of short acting Octreotide for up to 6 weeks in order to obtain an OctreoScan®, provided the patient returns to the Octreotide LAR fixed dose after the OctreoScan® has been obtained.
6. Confirmed presence of somatostatin receptors on all target lesions (for target/non-target/measurable lesions definition see §Appendix 2, Section 1 and 2, RECIST Criteria, Version 1.1) documented by CT/MRI scans, based on positive OctreoScan® imaging within 24 weeks prior to randomization in the study (to be centrally confirmed). The OctreoScan® should be one that was performed while the patient was on a fixed dose of Octreotide LAR. If a patient has had an OctreoScan® performed while Octreotide LAR treatment-naïve, the patient must have a repeat OctreoScan® performed after 3 months of Octreotide LAR treatments before entering the clinical study to prove that the index lesions or new lesions still meet the criteria for inclusion. It is acceptable to have patients temporarily switched to Octreotide s.c. (up to six weeks) in order to obtain an OctreoScan®, provided they return to the same fixed dose of Octreotide LAR prior to the scan.
7. The tumour uptake observed in each target lesion (for target/non-target/measurable lesions definition see §Appendix 2, Sections 1 and 2, RECIST Criteria, Version 1.1) using OctreoScan® must be ≥ normal liver uptake observed on planar imaging (to be centrally confirmed) (§Appendices 5 and 6).
8. Karnofsky Performance Score (KPS)>=60.
9. Presence of at least 1 measurable site of disease.
10. [Applicable only for France] All patients included in the trial must be affiliated with a social security regime or be a beneficiary of the same in order to be included in the study.

Exclusion Criteria:

1. Either serum creatinine >150 µmol/L (>1.7 mg/dL), or creatinine clearance <50 mL/min calculated by the Cockroft Gault method, eventually confirmed by measured creatinine clearance (or measured glomerular filtration rate (GFR) using plasma clearance methods, not gamma camera-based) <50 mL/min (the measured creatinine clearance / GFR is required only as confirmatory exam).
2. Hb concentration <5.0 mmol/L (<8.0 g/dL); WBC <2x109/L (2000/mm3); platelets <75x109/L (75x103/mm3).
3. Total bilirubin >3 x ULN.
4. Serum albumin <3.0 g/dL unless prothrombin time is within the normal range.
5. Pregnancy or lactation.
6. For female patients of childbearing potential (defined as < 2 years after last menstruation and not surgically sterile) and male patients, who are not surgically sterile or with female partners of childbearing potential: absence of effective, non-hormonal means of contraception (intrauterine contraceptive device, barrier method of contraception in conjunction with spermicidal gel) as defined in §Appendix 7.
7. Treatment with >30 mg Octreotide LAR at 3-4 weeks intervals within 12 weeks prior to randomization in the study.
8. Peptide receptor radionuclide therapy (PRRT) at any time prior to randomization in the study.
9. Any surgery, radioembolization, chemoembolization, chemotherapy and radiofrequency ablation within 12 weeks prior to randomization in the study.
10. Interferons, Everolimus (mTOR-inhibitors) or other systemic therapies within 4 weeks prior to randomization in the study.
11. Known brain metastases, unless these metastases have been treated and stabilized for at least 24 weeks, prior to enrollment in the study. Patients with a history of brain metastases must have a head CT with contrast to document stable disease prior to randomization in the study.
12. Uncontrolled congestive heart failure (NYHA II, III, IV).
13. Uncontrolled diabetes mellitus as defined by a fasting blood glucose >2 ULN.
14. Any patient receiving treatment with short-acting Octreotide, which cannot be interrupted for 24 h before and 24 h after the administration of 177Lu-DOTA0-Tyr3-Octreotate, or any patient receiving treatment with Octreotide LAR, which cannot be interrupted for at least 6 weeks before the administration of 177Lu-DOTA0-Tyr3-Octreotate, unless the tumour uptake on target lesions observed by OctreoScan® imaging during continued Octreotide LAR treatment is at least as high as normal liver uptake observed by planar imaging.
15. Patients with any other significant medical, psychiatric, or surgical condition, currently uncontrolled by treatment, which may interfere with the completion of the study.
16. Prior external beam radiation therapy to more than 25% of the bone marrow.
17. Current spontaneous urinary incontinence.
18. Other known co-existing malignancies except non-melanoma skin cancer and carcinoma in situ of the uterine cervix, unless definitively treated and proven no evidence of recurrence for 5 years.
19. Patients who have not provided a signed informed consent form to participate in the study, obtained prior to the start of any protocol related activities.
20. Patient with known incompatibility to CT Scans with I.V. contrast due to allergic reaction or renal insufficiency. If such a patient can be imaged with MRI, then the patient would not be excluded.
21. Patients who have participated in any therapeutic clinical study/received any investigational agent within the last 30 days are excluded from participation in this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 231 (Actual)
Dates: Start 2012-09-06 (Actual); Primary Completion 2015-07-31 (Actual); Study Completion 2021-01-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (39):
- United States (13):
  - Cedars-Sinai Medical Center Samuel Oschin Cancer Center, Los Angeles, California
  - Stanford Cancer Center, Palo Alto, California
  - Moffitt Cancer Center, Tampa, Florida
  - Northwestern Medical Faculty Foundation, Chicago, Illinois
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Duke University Medical Center, Durham, North Carolina
  - Kettering Medical Center, Kettering, Ohio
  - Perelman Center for Advanced Medicine, Philadelphia, Pennsylvania
  - Henry-Joyce Cancer Clinic, Nashville, Tennessee
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - Excel Diagnostics and Nuclear Oncology Center, Houston, Texas
- Digestive Oncology, Leuven Cancer Institute, Leuven, Brabant Flamand, Belgium
- France (6):
  - Centre Hospitalier Lyon-Sud, Lyon, Auvergne-Rhône-Alpes
  - Institut Claudius Regaud, Toulouse, Midi-Pyrénées
  - Hotel Dieu/CHU Nantes, Nantes, Pays de la Loire Region
  - Hôpital la Timone /CHU Marseille, Marseille, Provence-Alpes-Côte d'Azur Region
  - Hôpital Beaujon AP-HP, Clichy
  - Institut Gustave Roussy, Villejuif, Île-de-France Region
- Germany (4):
  - Klinikum Rechts Isar, Nuclear Medicine, Munich, Bavaria
  - Universitätsmedizin Mainz, Medizinische Klinik I Schwerpunkt Endokrinologie, Mainz, Rhineland-Palatinate
  - Zentralklinik Bad Berka, Bad Berka, Thuringia
  - Charité, Virchow-Klinikum, Gastroentrology, Hepatology & Endocrinology, Berlin
- Italy (6):
  - Istituto Oncologico Romagnolo per lo Studio dei Tumori, Meldola, Emilia-Romagna
  - IEO Istituto Europeo di Oncologia, Milan, Lombardy
  - Presidio Osp. Di Macerata, Macerata, The Marches
  - Azienda Ospedaliero - Universitaria Pisana (Presidio Ospedaliero S. Chiara), Pisa, Tuscany
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan
  - Università "Sapienza" di Roma, Facoltà di Medicina e Psicologia, Ospedale S. Andrea-Roma, Roma
- Portugal (2):
  - Centro Hospitalar e Universitario de Coimbra, Coimbra, Centro
  - Instituto Português de Oncologia, Porto, Norte
- Spain (2):
  - University Hospital of Bellvitge, Hospitalet de Llobregat (Barcelona), Catalonia
  - Ramon y Cajal University Hospital, Madrid
- United Kingdom (5):
  - University of Oxford, Oxford, South East England
  - Beatson Oncology Centre, Glasgow
  - Royal Free Hospital, London
  - Imperial College Healthcare Trust, Hammersmith Hospital, London
  - The Christie NHS foundation Trust, Manchester

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Strosberg JR, Caplin ME, Kunz PL, Ruszniewski PB, Bodei L, Hendifar A, Mittra E, Wolin EM, Yao JC, Pavel ME, Grande E, Van Cutsem E, Seregni E, Duarte H, Gericke G, Bartalotta A, Mariani MF, Demange A, Mutevelic S, Krenning EP; NETTER-1 investigators. 177Lu-Dotatate plus long-acting octreotide versus high-dose long-acting octreotide in patients with midgut neuroendocrine tumours (NETTER-1): final overall survival and long-term safety results from an open-label, randomised, controlled, phase 3 trial. Lancet Oncol. 2021 Dec;22(12):1752-1763. doi: 10.1016/S1470-2045(21)00572-6. Epub 2021 Nov 15. PMID 34793718
- [Derived] Strosberg J, Kunz PL, Hendifar A, Yao J, Bushnell D, Kulke MH, Baum RP, Caplin M, Ruszniewski P, Delpassand E, Hobday T, Verslype C, Benson A, Srirajaskanthan R, Pavel M, Mora J, Berlin J, Grande E, Reed N, Seregni E, Paganelli G, Severi S, Morse M, Metz DC, Ansquer C, Courbon F, Al-Nahhas A, Baudin E, Giammarile F, Taieb D, Mittra E, Wolin E, O'Dorisio TM, Lebtahi R, Deroose CM, Grana CM, Bodei L, Oberg K, Polack BD, He B, Mariani MF, Gericke G, Santoro P, Erion JL, Ravasi L, Krenning E; NETTER-1 study group. Impact of liver tumour burden, alkaline phosphatase elevation, and target lesion size on treatment outcomes with 177Lu-Dotatate: an analysis of the NETTER-1 study. Eur J Nucl Med Mol Imaging. 2020 Sep;47(10):2372-2382. doi: 10.1007/s00259-020-04709-x. Epub 2020 Mar 2. PMID 32123969
- [Derived] Strosberg J, Wolin E, Chasen B, Kulke M, Bushnell D, Caplin M, Baum RP, Kunz P, Hobday T, Hendifar A, Oberg K, Sierra ML, Thevenet T, Margalet I, Ruszniewski P, Krenning E; NETTER-1 Study Group. Health-Related Quality of Life in Patients With Progressive Midgut Neuroendocrine Tumors Treated With 177Lu-Dotatate in the Phase III NETTER-1 Trial. J Clin Oncol. 2018 Sep 1;36(25):2578-2584. doi: 10.1200/JCO.2018.78.5865. Epub 2018 Jun 7. PMID 29878866
- [Derived] Strosberg J, El-Haddad G, Wolin E, Hendifar A, Yao J, Chasen B, Mittra E, Kunz PL, Kulke MH, Jacene H, Bushnell D, O'Dorisio TM, Baum RP, Kulkarni HR, Caplin M, Lebtahi R, Hobday T, Delpassand E, Van Cutsem E, Benson A, Srirajaskanthan R, Pavel M, Mora J, Berlin J, Grande E, Reed N, Seregni E, Oberg K, Lopera Sierra M, Santoro P, Thevenet T, Erion JL, Ruszniewski P, Kwekkeboom D, Krenning E; NETTER-1 Trial Investigators. Phase 3 Trial of 177Lu-Dotatate for Midgut Neuroendocrine Tumors. N Engl J Med. 2017 Jan 12;376(2):125-135. doi: 10.1056/NEJMoa1607427. PMID 28076709
- See also: Health-Related Quality of Life in Patients With Progressive Midgut Neuroendocrine Tumors Treated With 177 Lu-Dotatate in the Phase III NETTER-1 Trial (J Clin Oncol . 2018 Sep 1;36(25):2578-2584) — https://pubmed.ncbi.nlm.nih.gov/29878866

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in 41 sites across 8 countries.
Period: Treatment Period
Arm/Group | 177Lu-DOTA0-Tyr3-Octreotate | Octreotide LAR
Started (All patients who received a randomization number, regardless of receiving study medication were included in the Randomized Set) | 117 | 114
Full Analysis Set (FAS) (All randomized participant were analyzed according to randomized treatment, regardless of the actual treatment received.) | 117 | 114
Safety Analysis Set (SAF) (All randomized patients who received at least one dose of active study medication. In the SAF, patients were analyzed based on actual treatment received.) | 111 | 112
FAS-Entered Long-term Follow-up | 101 | 99
Completed (refers to completion of a minimum of 72 weeks of treatment.) | 50 | 13
Not Completed | 67 | 101
Not completed — Progressive Disease | 19 | 64
Not completed — Physician Decision | 17 | 17
Not completed — Adverse Event | 13 | 10
Not completed — Non-compliance | 2 | 0
Not completed — Withdrawal by Subject | 10 | 9
Not completed — Other | 6 | 1
Period: Long-term Follow-Up Period
Arm/Group | 177Lu-DOTA0-Tyr3-Octreotate | Octreotide LAR
Started | 101 (FAS-Entered long-term follow-up) | 99 (FAS-Entered long-term follow-up)
Completed (Study ended 5 years from randomization of last participant or 158 deaths in the study achieved) | 24 | 19
Not Completed | 77 | 80
Not completed — Death | 69 | 64
Not completed — Consent withdrawal | 4 | 10
Not completed — Lost to Follow-up | 2 | 4
Not completed — Other | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 177Lu-DOTA0-Tyr3-Octreotate | Octreotide LAR | Total
Number analyzed (Participants) | 117 | 114 | 231
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.4 (9.34) | 64.0 (9.80) | 63.7 (9.55)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54 | 60 | 114
  Male | 63 | 54 | 117
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 1 | 0 | 1
  Black or African American | 5 | 5 | 10
  Hispanic | 6 | 3 | 9
  White | 93 | 96 | 189
  Other | 0 | 1 | 1
  Not Applicable | 12 | 9 | 21

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: Progression Free Survival (PFS) was defined as the time from randomization to documented centrally assessed disease progression, as evaluated by the Independent Review Committee (IRC), or death due to any cause. If a participant had no centrally assessed progression and had not died at the time of the primary endpoint analysis, the participant was regarded as censored in the context of a time to event analysis at the date of last evaluable tumor assessment. Disease progression was determined by objective tumor response status using Response Evaluation Criteria in Solid Tumors Criteria (RECIST v1.1).
Time Frame: From date of randomization until date of radiographic progression or date of death from any cause, whichever comes first until Primary Analysis cutoff date reached on 24July2015, assessed up to approximately 34 months
Population: Full Analysis Set (FAS).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | 177Lu-DOTA0-Tyr3-Octreotate | Octreotide LAR
Number analyzed (Participants) | 117 | 114
months | NA [NA to NA] — NA: not estimable due to number of censored participants at the time the analysis cut off date was reached. | 8.5 [5.8 to 9.1]
Statistical Analysis 1: Comparison: 177Lu-DOTA0-Tyr3-Octreotate vs Octreotide LAR; Test type: Superiority; p < 0.0001, Log Rank — Derived from a two-sided test between the two groups; Hazard Ratio (HR) = 0.177, 95% CI 2-sided [0.108 to 0.289] — Hazard ratio is expressed as Lu-DOTA-Tyr-Octreotate / Octreotide LAR and estimated from the corresponding Cox model

2. Secondary Outcome: Objective Response Rate (ORR)
Description: Objective Response Rate (ORR) was calculated as the proportion of patients with tumour size reduction (sum of partial responses (PR) and complete responses (CR)) according to RECIST 1.1.
Time Frame: From date of randomization until date of progression or date of death from any cause, whichever comes first until Primary Analysis cutoff date reached on 24July2015, assessed up to approximately 34 months
Population: Full Analysis Set (FAS). Only participants with available post-baseline CT scans were considered.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | 177Lu-DOTA0-Tyr3-Octreotate | Octreotide LAR
Number analyzed (Participants) | 102 | 100
Percentage of Participants | 14.7 [7.8 to 21.6] | 4.0 [0.2 to 7.8]
Statistical Analysis 1: Comparison: 177Lu-DOTA0-Tyr3-Octreotate vs Octreotide LAR; Test type: Superiority; p = 0.0141, Fisher Exact

3. Secondary Outcome: Overall Survival (OS)
Description: Overall Survival (OS) was defined as the time from the date of randomization to the date of death due to any cause or the date of last contact (censored observation) prior to the date of the data cut-off, and during the entire study period (i.e. the treatment period plus follow-up).
Time Frame: From date of randomization until date of death from any cause up to final safety cut-off date reached on 18Jan2021, assessed up to approximately 100 months
Population: Full Analysis Set (FAS).
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | 177Lu-DOTA0-Tyr3-Octreotate | Octreotide LAR
Number analyzed (Participants) | 117 | 114
Months | 48.0 [37.4 to 55.2] | 36.3 [25.9 to 51.7]
Statistical Analysis 1: Comparison: 177Lu-DOTA0-Tyr3-Octreotate vs Octreotide LAR; Test type: Superiority; p = 0.3039, Log Rank; Hazard Ratio (HR) = 0.84, 95% CI 2-sided [0.60 to 1.17]

4. Secondary Outcome: Rate of Overall Survival (OS)
Description: Survival estimates were collected every 12 Months up to 60 Months to compare OS between the two treatment groups.
Time Frame: 12 months, 24 months, 36 months, 48 months, 60 months
Population: Full Analysis Set (FAS).
Measure: Number (95% Confidence Interval); unit: Percentage of Survival Estimates
Arm/Group | 177Lu-DOTA0-Tyr3-Octreotate | Octreotide LAR
Number analyzed (Participants) | 117 | 114
Percentage of Survival Estimates
  12 months | 91.0 [84.0 to 95.1] | 79.7 [70.8 to 86.1]
  24 months | 76.0 [66.7 to 83.0] | 62.7 [52.6 to 71.2]
  36 months | 61.4 [51.4 to 69.9] | 50.1 [40.0 to 59.4]
  48 months | 49.5 [39.5 to 58.6] | 41.8 [31.8 to 51.4]
  60 months | 37.1 [27.8 to 46.4] | 35.4 [25.7 to 45.2]
Statistical Analysis 1: Comparison: 177Lu-DOTA0-Tyr3-Octreotate vs Octreotide LAR; Test type: Superiority; p = 0.3039, Log Rank; Cox Proportional Hazard = 0.84, 95% CI 2-sided [0.60 to 1.17] — Hazard Ratio of Lu-DOTA-Tyr-Octreotate vs. Octreotide LAR

5. Secondary Outcome: Time to Tumour Progression (TTP)
Description: Time to Tumour Progression (TTP) was defined as the time from randomization to progression centrally assessed. It included patients who dropped out due to toxicity, but omitted patients who died without measured progression (censored to last follow-up date or death date).
Time Frame: as for outcome 2
Population: Full Analysis Set (FAS).
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | 177Lu-DOTA0-Tyr3-Octreotate | Octreotide LAR
Number analyzed (Participants) | 117 | 114
Months | NA [NA to NA] — NA: not estimable due to number of censored participants at the time the analysis cut off date was reached. | 8.7 [6.0 to 11.1]
Statistical Analysis 1: Comparison: 177Lu-DOTA0-Tyr3-Octreotate vs Octreotide LAR; Test type: Superiority; p < 0.0001, Log Rank; Hazard Ratio (HR) = 0.137, 95% CI 2-sided [0.077 to 0.242]

6. Secondary Outcome: Duration of Response (DoR)
Description: The Duration of Response (DoR) was defined as the time from initially meeting the criteria for response (CR or PR) until the time of progression by RECIST 1.1.
Time Frame: as for outcome 2
Population: Full Analysis Set (FAS). Only Participants with an Objective Response are included in the analysis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | 177Lu-DOTA0-Tyr3-Octreotate | Octreotide LAR
Number analyzed (Participants) | 15 | 4
Months | NA [2.8 to NA] — NA: not estimable due to number of censored participants at the time the analysis cut off date was reached. | 1.9 [1.9 to NA] — NA: not estimable due to number of censored participants at the time the analysis cut off date was reached.

7. Secondary Outcome: Number of Participants With Adverse Events
Description: The distribution of adverse events was done via the analysis of frequencies for Adverse Event (AEs), Serious Adverse Event (SAEs) and Deaths, through the monitoring of relevant clinical and laboratory safety parameters.
Time Frame: From informed consent signature through study completion reached at final safety cutoff date on 18July2021, assessed up to approximately 101 Months
Population: Safety Analysis Set (SAF).
Measure: Count of Participants; unit: Participants
Arm/Group | 177Lu-DOTA0-Tyr3-Octreotate | Octreotide LAR
Number analyzed (Participants) | 111 | 112
Participants
  Adverse Events (AEs) | 105 | 90
  Serious Adverse Events (SAEs) | 40 | 31
  Deaths during treatment period | 4 | 5
  Deaths during follow-up period | 66 | 63

8. Secondary Outcome: Change From Baseline in the EORTC QLQ-C30 Questionnaire
Description: The Quality of Life Questionnaire C30 (QLQ-C30) was developed by the European Organization for Research and Treatment of Cancer (EORTC) to assess quality of life in cancer patients. It includes five function domains (physical, emotional, social, role, cognitive), eight symptoms (fatigue, pain, nausea/vomiting, constipation, diarrhea, insomnia, dyspnea, and appetite loss), as well as global health/quality-of-life and financial impact. Subjects respond on a four-point scale from "not at all" to "very much" for most items. Raw scores are linearly transformed so each score ranged a 0-100, where higher scores indicate worse symptoms (e.g., more severe/worsened) and lower scores indicate less symptoms (e.g., less severe/improvement).
Time Frame: Inclusion (Baseline) (BL), Week 72, Week 120
Population: Safety Analysis Set (SAF). Values at Inclusion were taken from last non-missing value prior to randomization (the only scheduled pre-randomization assessment was at the Baseline visit). Calculations at each visit included only participants with scores at the visit and Inclusion.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | 177Lu-DOTA0-Tyr3-Octreotate | Octreotide LAR
Number analyzed (Participants) | 111 | 112
Scores on a scale
  Physical functioning: chg from BL @ wk 72 (n=33,11): number analyzed (Participants) | 33 | 11
  Physical functioning: chg from BL @ wk 72 (n=33,11) | 3.232 (12.4857) | -4.242 (10.0101)
  Physical functioning: chg from BL @ wk 120 (n=2,0): number analyzed (Participants) | 2 | 0
  Physical functioning: chg from BL @ wk 120 (n=2,0) | -3.333 (4.7140) |
  Role functioning: chg from BL @ wk 72 (n=33,11): number analyzed (Participants) | 33 | 11
  Role functioning: chg from BL @ wk 72 (n=33,11) | 5.051 (33.1989) | -3.030 (16.3608)
  Role functioning: chg from BL @ wk 120 (n=2,0): number analyzed (Participants) | 2 | 0
  Role functioning: chg from BL @ wk 120 (n=2,0) | 8.333 (11.7851) |
  Emotional functioning: chg from BL @ wk 72 (n=33,11): number analyzed (Participants) | 33 | 11
  Emotional functioning: chg from BL @ wk 72 (n=33,11) | 7.744 (22.6602) | 6.061 (17.9083)
  Emotional functioning: chg from BL @ wk 120 (n=2,0): number analyzed (Participants) | 2 | 0
  Emotional functioning: chg from BL @ wk 120 (n=2,0) | 12.500 (5.8926) |
  Cognitive functioning: chg from BL @ wk 72 (n=33,11): number analyzed (Participants) | 33 | 11
  Cognitive functioning: chg from BL @ wk 72 (n=33,11) | 5.556 (15.9571) | 1.515 (13.8535)
  Cognitive functioning: chg from BL @ wk 120 (n=2,0): number analyzed (Participants) | 2 | 0
  Cognitive functioning: chg from BL @ wk 120 (n=2,0) | 16.667 (23.5702) |
  Social functioning: chg from BL @ wk 72 (n=33,11): number analyzed (Participants) | 33 | 11
  Social functioning: chg from BL @ wk 72 (n=33,11) | 8.586 (28.9039) | -7.576 (18.8025)
  Social functioning: chg from BL @ wk 120 (n=2,0): number analyzed (Participants) | 2 | 0
  Social functioning: chg from BL @ wk 120 (n=2,0) | 8.333 (35.3553) |
  Global Health Status/QoL: chg from BL @ wk 72 (n=33,11): number analyzed (Participants) | 33 | 11
  Global Health Status/QoL: chg from BL @ wk 72 (n=33,11) | 5.556 (21.4155) | 1.515 (10.4205)
  Global Health Status/QoL: chg from BL @ wk 120 (n=2,0): number analyzed (Participants) | 2 | 0
  Global Health Status/QoL: chg from BL @ wk 120 (n=2,0) | -16.667 (0.0000) |
  Fatigue: chg from BL @ wk 72 (n=33,11): number analyzed (Participants) | 33 | 11
  Fatigue: chg from BL @ wk 72 (n=33,11) | -7.239 (24.7084) | -2.020 (13.8939)
  Fatigue: chg from BL @ wk 120 (n=2,0): number analyzed (Participants) | 2 | 0
  Fatigue: chg from BL @ wk 120 (n=2,0) | 11.111 (0.0000) |
  Nausea & Vomiting: chg from BL @ wk 72 (n=33,11): number analyzed (Participants) | 33 | 11
  Nausea & Vomiting: chg from BL @ wk 72 (n=33,11) | -4.545 (15.1799) | -4.545 (7.7850)
  Nausea & Vomiting: chg from BL @ wk 120 (n=2,0): number analyzed (Participants) | 2 | 0
  Nausea & Vomiting: chg from BL @ wk 120 (n=2,0) | 0.000 (0.0000) |
  Pain: chg from BL @ wk 72 (n=33,11): number analyzed (Participants) | 33 | 11
  Pain: chg from BL @ wk 72 (n=33,11) | -8.586 (22.4850) | -3.030 (10.0504)
  Pain: chg from BL @ wk 120 (n=2,0): number analyzed (Participants) | 2 | 0
  Pain: chg from BL @ wk 120 (n=2,0) | 0.000 (23.5702) |
  Dyspnoea: chg from BL @ wk 72 (n=33,11): number analyzed (Participants) | 33 | 11
  Dyspnoea: chg from BL @ wk 72 (n=33,11) | -3.030 (22.6134) | 3.030 (27.7070)
  Dyspnoea: chg from BL @ wk 120 (n=2,0): number analyzed (Participants) | 2 | 0
  Dyspnoea: chg from BL @ wk 120 (n=2,0) | 0.000 (0.0000) |
  Insomnia: chg from BL @ wk 72 (n=33,11): number analyzed (Participants) | 33 | 11
  Insomnia: chg from BL @ wk 72 (n=33,11) | 0.000 (26.3523) | 6.061 (29.1288)
  Insomnia: chg from BL @ wk 120 (n=2,0): number analyzed (Participants) | 2 | 0
  Insomnia: chg from BL @ wk 120 (n=2,0) | 33.333 (47.1405) |
  Appetite loss: chg from BL @ wk 72 (n=33,11): number analyzed (Participants) | 33 | 11
  Appetite loss: chg from BL @ wk 72 (n=33,11) | -8.081 (20.4639) | 9.091 (21.5557)
  Appetite loss: chg from BL @ wk 120 (n=2,0): number analyzed (Participants) | 2 | 0
  Appetite loss: chg from BL @ wk 120 (n=2,0) | 0.000 (0.0000) |
  Constipation: chg from BL @ wk 72 (n=33,11): number analyzed (Participants) | 33 | 11
  Constipation: chg from BL @ wk 72 (n=33,11) | 0.000 (18.6339) | 0.000 (14.9071)
  Constipation: chg from BL @ wk 120 (n=2,0): number analyzed (Participants) | 2 | 0
  Constipation: chg from BL @ wk 120 (n=2,0) | 0.000 (0.0000) |
  Diarrhoea: chg from BL @ wk 72 (n=33,11): number analyzed (Participants) | 33 | 11
  Diarrhoea: chg from BL @ wk 72 (n=33,11) | -12.121 (36.1499) | -3.030 (27.7070)
  Diarrhoea: chg from BL @ wk 120 (n=2,0): number analyzed (Participants) | 2 | 0
  Diarrhoea: chg from BL @ wk 120 (n=2,0) | -16.667 (23.5702) |
  Financial difficulties: chg from BL @ wk 72 (n=33,11): number analyzed (Participants) | 33 | 11
  Financial difficulties: chg from BL @ wk 72 (n=33,11) | -7.071 (33.0798) | 6.061 (20.1008)
  Financial difficulties: chg from BL @ wk 120 (n=2,0): number analyzed (Participants) | 2 | 0
  Financial difficulties: chg from BL @ wk 120 (n=2,0) | -16.667 (70.7107) |

9. Secondary Outcome: Change From Baseline in the EORTC Quality of Life Questionnaire - Neuroendocrine Carcinoid Module (EORTC QLQ-GINET21)
Description: The Quality of Life GI Neuroendocrine Tumor survey (QLQ GINET21) contains a total of 21 items: four single-item assessments relating to muscle and/or bone pain (MBP), body image (BI), information (INF) and sexual functioning (SX), together with 17 items organized into five proposed scales: endocrine symptoms (ED; three items), GI symptoms (GI; five items), treatment-related symptoms (TR; three items), social functioning (SF) and disease-related worries (DRW; three items). The response format of the questionnaire is a four-point Likert scale. Responses are linearly transformed to a 0-100 scale using EORTC guidelines, with higher scores reflecting more severe symptoms.
Time Frame: Inclusion (Baseline) (BL), Week 72, Week 120
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | 177Lu-DOTA0-Tyr3-Octreotate | Octreotide LAR
Number analyzed (Participants) | 112 | 111
Scores on a scale
  Endocrine scale: chg from BL @ wk 72 (n=33,11): number analyzed (Participants) | 33 | 11
  Endocrine scale: chg from BL @ wk 72 (n=33,11) | -8.754 (20.1762) | -11.111 (21.0819)
  Endocrine scale: chg from BL @ wk 120 (n=2,0): number analyzed (Participants) | 2 | 0
  Endocrine scale: chg from BL @ wk 120 (n=2,0) | 0.000 (0.0000) |
  G.I. scale: chg from BL @ wk 72 (n=33,11): number analyzed (Participants) | 33 | 11
  G.I. scale: chg from BL @ wk 72 (n=33,11) | -2.727 (15.3083) | 2.424 (10.0101)
  G.I. scale: chg from BL @ wk 120 (n=2,0): number analyzed (Participants) | 2 | 0
  G.I. scale: chg from BL @ wk 120 (n=2,0) | -13.333 (0.0000) |
  Treatment scale: chg from BL @ wk 72 (n=21,5): number analyzed (Participants) | 21 | 5
  Treatment scale: chg from BL @ wk 72 (n=21,5) | -8.995 (14.9563) | 0.000 (11.1111)
  Treatment scale: chg from BL @ wk 120 (n=1,0): number analyzed (Participants) | 1 | 0
  Treatment scale: chg from BL @ wk 120 (n=1,0) | -16.667 (NA) — Only one participant analyzed |
  Social function scale: chg from BL @ wk 72 (n=33,11): number analyzed (Participants) | 33 | 11
  Social function scale: chg from BL @ wk 72 (n=33,11) | -7.576 (23.3985) | -7.576 (21.1217)
  Social function scale: chg from BL @ wk 120 (n=2,0): number analyzed (Participants) | 2 | 0
  Social function scale: chg from BL @ wk 120 (n=2,0) | 11.111 (0.0000) |
  Diseases rel. worries scale: chg from BL @ wk 72 (n=33,11): number analyzed (Participants) | 33 | 11
  Diseases rel. worries scale: chg from BL @ wk 72 (n=33,11) | -6.061 (27.9289) | 1.010 (33.7765)
  Diseases rel. worries scale: chg from BL @ wk 120 (n=2,0): number analyzed (Participants) | 2 | 0
  Diseases rel. worries scale: chg from BL @ wk 120 (n=2,0) | 33.333 (31.4270) |
  Muscle/Bone pain symptom: chg from BL @ wk 72 (n=33,10): number analyzed (Participants) | 33 | 10
  Muscle/Bone pain symptom: chg from BL @ wk 72 (n=33,10) | -5.051 (33.4594) | -16.667 (36.0041)
  Muscle/Bone pain symptom: chg from BL @ wk 120 (n=2,0): number analyzed (Participants) | 2 | 0
  Muscle/Bone pain symptom: chg from BL @ wk 120 (n=2,0) | -16.667 (23.5702) |
  Sexual function: chg from BL @ wk 72 (n=21,7): number analyzed (Participants) | 21 | 7
  Sexual function: chg from BL @ wk 72 (n=21,7) | 6.349 (40.3031) | 14.286 (17.8174)
  Sexual function: chg from BL @ wk 120 (n=2,0): number analyzed (Participants) | 2 | 0
  Sexual function: chg from BL @ wk 120 (n=2,0) | 50.000 (70.7107) |
  Information/Communication: chg from BL @ wk 72 (n=33,11): number analyzed (Participants) | 33 | 11
  Information/Communication: chg from BL @ wk 72 (n=33,11) | -4.040 (26.0309) | -12.121 (30.8139)
  Information/Communication: chg from BL @ wk 120 (n=2,0): number analyzed (Participants) | 2 | 0
  Information/Communication: chg from BL @ wk 120 (n=2,0) | 0.000 (0.0000) |
  Body image: chg from BL @ wk 72 (n=33,11): number analyzed (Participants) | 33 | 11
  Body image: chg from BL @ wk 72 (n=33,11) | -4.040 (18.1766) | -3.030 (17.9787)
  Body image: chg from BL @ wk 120 (n=2,0): number analyzed (Participants) | 2 | 0
  Body image: chg from BL @ wk 120 (n=2,0) | 16.667 (23.5702) |

ADVERSE EVENTS:
Time Frame: From informed consent signature through study completion reached at final safety cutoff date on 18July2021, assessed up to approximately 101 Months.
Description: Any sign or symptom that occurs after written informed consent provided.
Arm/Group | 177Lu-DOTA0-Tyr3-Octreotate | Octreotide LAR
All-Cause Mortality (participants affected / at risk) | 70/111 | 68/112
Serious Adverse Events (participants affected / at risk) | 40/111 | 31/112
Other Adverse Events (participants affected / at risk) | 105/111 | 90/112
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 177Lu-DOTA0-Tyr3-Octreotate (N=111) | Octreotide LAR (N=112)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Lymphopenia (Blood and lymphatic system disorders) | 2 | 0
Myelodysplastic syndrome (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Refractory cytopenia with unilineage dysplasia (Blood and lymphatic system disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 1 | 0
Arteriospasm coronary (Cardiac disorders) | 0 | 1
Atrioventricular block second degree (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Silent myocardial infarction (Cardiac disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 3 | 1
Abdominal pain lower (Gastrointestinal disorders) | 0 | 2
Anal haemorrhage (Gastrointestinal disorders) | 0 | 1
Ascites (Gastrointestinal disorders) | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Duodenal obstruction (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 0
Gastrointestinal obstruction (Gastrointestinal disorders) | 0 | 1
Haematochezia (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 1
Impaired gastric emptying (Gastrointestinal disorders) | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Malignant bowel obstruction (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 2
Vomiting (Gastrointestinal disorders) | 2 | 2
Complication of device insertion (General disorders) | 1 | 0
Device occlusion (General disorders) | 1 | 0
General physical health deterioration (General disorders) | 2 | 2
Generalised oedema (General disorders) | 0 | 1
Injection site hypersensitivity (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
Cholestasis (Hepatobiliary disorders) | 1 | 0
Hepatic encephalopathy (Hepatobiliary disorders) | 1 | 0
Hepatocellular injury (Hepatobiliary disorders) | 1 | 0
Clostridium difficile infection (Infections and infestations) | 1 | 0
Device related infection (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 1 | 0
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 2 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 1
Limb traumatic amputation (Injury, poisoning and procedural complications) | 1 | 0
Procedural complication (Injury, poisoning and procedural complications) | 1 | 0
Blood creatinine increased (Investigations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 1
Fluid retention (Metabolism and nutrition disorders) | 1 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Carcinoid crisis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 5
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Refractory cytopenia with multilineage dysplasia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tumour invasion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Thrombotic cerebral infarction (Nervous system disorders) | 0 | 1
Transient global amnesia (Nervous system disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 0
Delirium (Psychiatric disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 4 | 1
Acute prerenal failure (Renal and urinary disorders) | 1 | 0
Renal impairment (Renal and urinary disorders) | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Coronary artery bypass (Surgical and medical procedures) | 1 | 0
Inferior vena cava syndrome (Vascular disorders) | 1 | 0
Pulmonary embolism (Vascular disorders) | 1 | 0
Shock (Vascular disorders) | 1 | 0
Syncope (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 177Lu-DOTA0-Tyr3-Octreotate (N=111) | Octreotide LAR (N=112)
Anaemia (Blood and lymphatic system disorders) | 18 | 8
Lymphopenia (Blood and lymphatic system disorders) | 18 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 16 | 0
Palpitations (Cardiac disorders) | 6 | 6
Abdominal distension (Gastrointestinal disorders) | 18 | 14
Abdominal pain (Gastrointestinal disorders) | 28 | 21
Abdominal pain upper (Gastrointestinal disorders) | 6 | 2
Constipation (Gastrointestinal disorders) | 11 | 6
Diarrhoea (Gastrointestinal disorders) | 32 | 20
Dyspepsia (Gastrointestinal disorders) | 7 | 7
Flatulence (Gastrointestinal disorders) | 7 | 6
Nausea (Gastrointestinal disorders) | 74 | 13
Vomiting (Gastrointestinal disorders) | 59 | 9
Asthenia (General disorders) | 9 | 8
Fatigue (General disorders) | 43 | 30
Influenza like illness (General disorders) | 6 | 4
Oedema peripheral (General disorders) | 18 | 10
Pyrexia (General disorders) | 8 | 3
Urinary tract infection (Infections and infestations) | 7 | 7
Alanine aminotransferase increased (Investigations) | 7 | 7
Aspartate aminotransferase increased (Investigations) | 5 | 8
Blood alkaline phosphatase increased (Investigations) | 7 | 8
Blood bilirubin increased (Investigations) | 7 | 3
Blood creatinine increased (Investigations) | 7 | 6
Gamma-glutamyltransferase increased (Investigations) | 7 | 9
Lymphocyte count decreased (Investigations) | 12 | 2
Platelet count decreased (Investigations) | 13 | 2
Weight decreased (Investigations) | 9 | 8
White blood cell count decreased (Investigations) | 7 | 1
Decreased appetite (Metabolism and nutrition disorders) | 24 | 12
Hyperglycaemia (Metabolism and nutrition disorders) | 11 | 10
Hypokalaemia (Metabolism and nutrition disorders) | 9 | 10
Hyponatraemia (Metabolism and nutrition disorders) | 7 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 12 | 11
Back pain (Musculoskeletal and connective tissue disorders) | 15 | 11
Muscle spasms (Musculoskeletal and connective tissue disorders) | 7 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 5 | 6
Pain in extremity (Musculoskeletal and connective tissue disorders) | 12 | 6
Dizziness (Nervous system disorders) | 19 | 10
Dysgeusia (Nervous system disorders) | 9 | 2
Headache (Nervous system disorders) | 21 | 6
Syncope (Nervous system disorders) | 6 | 2
Anxiety (Psychiatric disorders) | 13 | 6
Insomnia (Psychiatric disorders) | 3 | 8
Haematuria (Renal and urinary disorders) | 7 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 12 | 8
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 12 | 9
Alopecia (Skin and subcutaneous tissue disorders) | 13 | 2
Flushing (Vascular disorders) | 16 | 10
Hypertension (Vascular disorders) | 13 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.